CLINICAL TRIAL: NCT05832996
Title: Randomized Controlled Study of Cooled Versus Room-Temperature Artificial Tears for Reducing Surface Irritation Following Intravitreal Injection
Brief Title: Cool vs Room-temperature Artificial Tears
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202201397
Record Dates: First submitted 2023-03-14; First posted 2023-04-27 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Retinopathy With Macular Edema of Both Eyes (Diagnosis); Central Retinal Vein Occlusion With Macular Edema; Exudative Age-Related Macular Degeneration, Unspecified Eye; Cystoid Macular Edema; Ocular Surface Disease; Dry Eye Sensation; Eye Pain
MeSH Terms: conditions — Disease; Macular Edema; Eye Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cooled artificial tear group (Experimental): Stored at 4 degree Celsius
  Interventions: Drug: Refresh Plus Preservative-free Lubricant Eye Drops
- Room temperature artificial tear group (Active Comparator): Stored at 25 degree Celsius
  Interventions: Drug: Refresh Plus Preservative-free Lubricant Eye Drops

INTERVENTIONS:
Drug: Refresh Plus Preservative-free Lubricant Eye Drops — Refresh Plus Preservative-free Lubricant Eye Drops at either 4 or 25 degree Celsius

SUMMARY:
Background and Objective: To evaluate the efficacy of cooled versus room temperature artificial tears in reducing post intravitreal injection (IVI) ocular discomfort.

Patients and Methods: Patients receiving IVI were randomized to either cooled or room temperature tears intervention groups. Both groups rated their ocular discomfort following IVI before intervention and again after administration of cooled or room temperature tears.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were receiving standard intravitreal injections for their exudative age-related macular degeneration, cystoid macular edema, diabetic macular edema, proliferative diabetic retinopathy, retinal vein occlusion with macular edema, or retinal neovascularization.

Exclusion Criteria:

* Inability or lack of willingness to participate in the study
* Active ocular infection including infectious uveitis
* First time receiving intravitreal injection
* Those who reported never having ocular discomfort following intravitreal injections on the pre-injection questionnaire
* Less than 18 years of age

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Jin, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics - Department of Ophthalmology, Iowa City, Iowa, United States

REFERENCES:
- [Background] Peyman GA, Lad EM, Moshfeghi DM. Intravitreal injection of therapeutic agents. Retina. 2009 Jul-Aug;29(7):875-912. doi: 10.1097/IAE.0b013e3181a94f01. PMID 19584648
- [Background] Patel SN, Gangaputra S, Sternberg P Jr, Kim SJ. Prophylaxis measures for postinjection endophthalmitis. Surv Ophthalmol. 2020 Jul-Aug;65(4):408-420. doi: 10.1016/j.survophthal.2019.12.005. Epub 2020 Jan 7. PMID 31923477
- [Background] Grzybowski A, Kanclerz P, Myers WG. The use of povidone-iodine in ophthalmology. Curr Opin Ophthalmol. 2018 Jan;29(1):19-32. doi: 10.1097/ICU.0000000000000437. PMID 28984794
- [Background] Swift W, Bair JA, Chen W, Li M, Lie S, Li D, Yang M, Shatos MA, Hodges RR, Kolko M, Utheim TP, Scott W, Dartt DA. Povidone iodine treatment is deleterious to human ocular surface conjunctival cells in culture. BMJ Open Ophthalmol. 2020 Sep 16;5(1):e000545. doi: 10.1136/bmjophth-2020-000545. eCollection 2020. PMID 32995498
- [Background] Saedon H, Nosek J, Phillips J, Narendran N, Yang YC. Ocular surface effects of repeated application of povidone iodine in patients receiving frequent intravitreal injections. Cutan Ocul Toxicol. 2017 Dec;36(4):343-346. doi: 10.1080/15569527.2017.1291665. Epub 2017 Feb 28. PMID 28166657
- [Background] Laude A, Lim JW, Srinagesh V, Tong L. The effect of intravitreal injections on dry eye, and proposed management strategies. Clin Ophthalmol. 2017 Aug 16;11:1491-1497. doi: 10.2147/OPTH.S136500. eCollection 2017. PMID 28860698
- [Background] Dohlman TH, Lertsuwanroj B, D'Amico DJ, Ciralsky JB, Kiss S. Evaluation of signs and symptoms of ocular surface disease after intravitreal injection. Acta Ophthalmol. 2019 Dec;97(8):e1154-e1156. doi: 10.1111/aos.14146. Epub 2019 Jun 25. No abstract available. PMID 31237739
- [Background] Segal O, Segal-Trivitz Y, Nemet AY, Cohen P, Geffen N, Mimouni M. Anxiety levels and perceived pain intensity during intravitreal injections. Acta Ophthalmol. 2016 Mar;94(2):203-4. doi: 10.1111/aos.12802. Epub 2015 Jul 28. No abstract available. PMID 26215781
- [Background] Chaturvedi R, Wannamaker KW, Riviere PJ, Khanani AM, Wykoff CC, Chao DL. Real-World Trends in Intravitreal Injection Practices among American Retina Specialists. Ophthalmol Retina. 2019 Aug;3(8):656-662. doi: 10.1016/j.oret.2019.03.023. Epub 2019 Apr 4. PMID 31133544
- [Background] Avery RL, Bakri SJ, Blumenkranz MS, Brucker AJ, Cunningham ET Jr, D'Amico DJ, Dugel PU, Flynn HW Jr, Freund KB, Haller JA, Jumper JM, Liebmann JM, McCannel CA, Mieler WF, Ta CN, Williams GA. Intravitreal injection technique and monitoring: updated guidelines of an expert panel. Retina. 2014 Dec;34 Suppl 12:S1-S18. doi: 10.1097/IAE.0000000000000399. PMID 25489719
- [Background] Kaplan RI, Drinkwater OJ, Lee RH, Chod RB, Barash A, Giovinazzo JV, Gologorsky D, Jansen ME, Rosen RB, Gentile RC. Pain Control after Intravitreal Injection Using Topical Nepafenac 0.3% or Pressure Patching: A Randomized, Placebo-Controlled Trial. Ophthalmol Retina. 2019 Oct;3(10):860-866. doi: 10.1016/j.oret.2019.04.022. Epub 2019 Apr 26. PMID 31221565
- [Background] Rifkin L, Schaal S. Shortening ocular pain duration following intravitreal injections. Eur J Ophthalmol. 2012 Nov-Dec;22(6):1008-12. doi: 10.5301/ejo.5000147. Epub 2012 Apr 24. PMID 22562296
- [Background] Gaynes BI, Fiscella R. Topical nonsteroidal anti-inflammatory drugs for ophthalmic use: a safety review. Drug Saf. 2002;25(4):233-50. doi: 10.2165/00002018-200225040-00002. PMID 11994027
- [Background] Fujishima H, Yagi Y, Shimazaki J, Tsubota K. Effects of artificial tear temperature on corneal sensation and subjective comfort. Cornea. 1997 Nov;16(6):630-4. PMID 9395871
- [Background] Hu Youwei J, Chang B. Effect of cooling proparacaine 0.5% eye drops on patient's comfort during instillation. Eye (Lond). 2015 Aug;29(8):1112-3. doi: 10.1038/eye.2015.59. Epub 2015 Apr 24. No abstract available. PMID 25907208
- [Background] Ramos MS, Xu LT, Singuri S, Castillo Tafur JC, Arepalli S, Ehlers JP, Kaiser PK, Singh RP, Rachitskaya AV, Srivastava SK, Sears JE, Schachat AP, Babiuch AS, Sharma S, Martin DF, Lowder CY, Singh AD, Yuan A, Nowacki AS. Patient-Reported Complications after Intravitreal Injection and Their Predictive Factors. Ophthalmol Retina. 2021 Jul;5(7):625-632. doi: 10.1016/j.oret.2020.09.024. Epub 2020 Oct 12. PMID 33059077
- [Background] Messmer EM. The pathophysiology, diagnosis, and treatment of dry eye disease. Dtsch Arztebl Int. 2015 Jan 30;112(5):71-81; quiz 82. doi: 10.3238/arztebl.2015.0071. PMID 25686388
- [Background] Bitton E, Crncich V, Brunet N. Does the temperature of an artificial tear affect its comfort? Clin Exp Optom. 2018 Sep;101(5):641-647. doi: 10.1111/cxo.12664. Epub 2018 Feb 18. PMID 29457271
- [Background] Pucker AD, Ng SM, Nichols JJ. Over the counter (OTC) artificial tear drops for dry eye syndrome. Cochrane Database Syst Rev. 2016 Feb 23;2:CD009729. doi: 10.1002/14651858.CD009729.pub2. PMID 26905373
- [Background] Walsh K, Jones L. The use of preservatives in dry eye drops. Clin Ophthalmol. 2019 Aug 1;13:1409-1425. doi: 10.2147/OPTH.S211611. eCollection 2019. PMID 31447543

RESULTS

PARTICIPANT FLOW:
Groups:
- Cooled Artificial Tear Group: Stored at 4 degree Celsius
  Refresh Plus Preservative-free Lubricant Eye Drops: Refresh Plus Preservative-free Lubricant Eye Drops at 4 degree Celsius
- Room Temperature Artificial Tear Group: Stored at 25 degree Celsius
  Refresh Plus Preservative-free Lubricant Eye Drops: Refresh Plus Preservative-free Lubricant Eye Drops at 4 degree Celsius
Period: Overall Study
Arm/Group | Cooled Artificial Tear Group | Room Temperature Artificial Tear Group
Started | 56 | 68
Completed | 48 | 61
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cooled Artificial Tear Group | Room Temperature Artificial Tear Group | Total
Number analyzed (Participants) | 48 | 61 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (15.9) | 68.3 (15.4) | 68.7 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 45 | 77
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 47 | 59 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Cooled Versus Room Temperature Artificial Tears in Reducing Post Intravitreal Injection Ocular Discomfort as Measured by Pain Scale Survey.
Description: The level of subjectively reported pain scale from 1 to 10, where 1 is minimal pain and 10 is extreme pain
Time Frame: with 72 hours of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cooled Artificial Tear Group | Room Temperature Artificial Tear Group
Number analyzed (Participants) | 48 | 61
score on a scale | 2.21 (0.2) | 1.95 (0.2)

ADVERSE EVENTS:
Time Frame: The specific period time over which adverse event data were collected was 4 months, which was the entire duration of the study
Groups:
- Room Temperature Artificial Tear Group: Stored at 25 degree Celsius
  Refresh Plus Preservative-free Lubricant Eye Drops: Refresh Plus Preservative-free Lubricant Eye Drops at 25 degree Celsius
Arm/Group | Cooled Artificial Tear Group | Room Temperature Artificial Tear Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/61
Other Adverse Events (participants affected / at risk) | 0/48 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT05832996/Prot_001.pdf
  • Informed Consent Form (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT05832996/ICF_003.pdf